CLINICAL TRIAL: NCT05355623
Title: Surgical Repair of Vaginal Wall Prolapse Using Gamma Irradiated Amniotic Membrane as a Scaffold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMGAD SAMEEH
Record Dates: First submitted 2022-04-19; First posted 2022-05-02 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Vaginal Wall Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Intervention Model Description: compare between the usage of Gamma irradiated sterilized amniotic membrane as a graft versus conventional classical repair in terms of: Effectiveness, symptoms relief, healing, and infection rate.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- amniotic membrane graft (Active Comparator): patients in which the surgical vaginal repair will be done with the application of a sterilized (gamma irradiated) amniotic membrane.
  Interventions: Procedure: Vaginal Repair
- surgical vaginal repair (Active Comparator): patients in which the surgical vaginal repair will be done without any graft.
  Interventions: Procedure: Vaginal Repair

INTERVENTIONS:
Procedure: Vaginal Repair — Vaginal Repair will be done either by application of sterilized (gamma irradiated) amniotic membrane or by Classical repair

SUMMARY:
The surgical repair of vaginal wall prolapse continues to remain one of the most difficult challenges in female pelvic floor reconstruction. The recurrence rate after standard colporrhaphy ranges from 40-60 %. This high recurrence rate creates the necessity for developing new surgical techniques and better long-term solutions. Surgeons have been investigating the use of synthetic and biological grafts in vaginal wall prolapse repairs

DETAILED DESCRIPTION:
The surgical repair of vaginal wall prolapse continues to remain one of the most difficult challenges in female pelvic floor reconstruction. The recurrence rate after standard colporrhaphy ranges from 40-60 %. This high recurrence rate creates the necessity for developing new surgical techniques and better long-term solutions. Surgeons have been investigating the use of synthetic and biological grafts in vaginal wall prolapse repairs. The use of an absorbable polyglactin 910 mesh (Vicryl) has shown little benefit in its use to correct vaginal wall prolapse (42%), and the use of a synthetic permanent polypropylene mesh for vaginal repair shows a mesh erosion rate of 18%, de novo urgency rate of 20%, and dyspareunia 22% postoperatively. The mesh erosion rate or infection rate increased four-fold when the mesh was introduced vaginally as compared to the abdominal route in pelvic floor reconstruction cases.

Many pelvic surgeons are now using biological grafts for vaginal prolapse surgery, such as cadaveric fascia lata, cadaveric dermis, porcine small intestine, porcine dermis, or bovine pericardium, which are not used in the Middle East for cultural reasons. A new skin tissue-generated matrix has given some hope but is expensive. The use of Amniotic Membrane came to our attention as a possible biological graft material, since it is non-immunogenic, it will not be rejected, and as of protein nature, will be integrated and absorbed by the body after attracting fibrin and collagen, giving necessary support.

Human amniotic membrane is a tough membrane derived from the fetal membranes. Human amniotic membrane is believed to be non-immunogenic, Antibodies or cell-mediated immune response to the amniotic membrane have not been demonstrated, suggesting low antigenicity and hence the recipient will not reject it. Therefore, the use of systemic immunosuppressive drugs is not required.

Some surgeons have described the use of fresh human amniotic membrane for transplantation, but it is not without the risk of infection.

Another important aspect that makes human amniotic epithelial cells (hAECs) and fetal membrane-derived stromal cells attractive for potential stem cell-based therapies is their low antigenicity. The hAECs also release several anti-inflammatory factors that lead to a significant reduction in HLA class II antigen-presenting cells found at sites of injury that prevent apoptosis, enhance wound healing and host cell proliferation, and suppress profibrotic transforming growth factor-beta isoforms and type II transforming growth factor-beta receptors in myofibroblast cells that deposit collagen, which leads to fibrosis. Amniotic membrane has diverse properties against bacterial and viral infections, stores antibiotics, and releases them over the course of a few days, and recently has been shown to produce potent natural antimicrobials. Clinical studies suggest that the amniotic membrane as a biologic dressing has 2 primary favorable effects in addition to being an anatomical barrier as it facilitates epithelialization by acting as a basement membrane substrate, facilitates migration of epithelial cells, reinforces adhesion of the basal epithelium, promotes cellular differentiation, and prevents cellular apoptosis, and it inhibits inflammation and fibrosis. Amnion graft, either fresh or dried, is a promising adjunctive procedure for decreasing the recurrence of adhesions and encouraging endometrial regeneration. Both grafts seem to be equally effective; however, dried amnion graft holds some advantages easy availability, prevention of cross-infection, and easier surgical application. The use of non sterilized amniotic membrane is supposed to increase the risk of fungal, bacterial, or viral diseases transmission from donors. The amniotic membrane graft is a natural human protein, attracting collagen formation, fibrinogen, and causing mild fibrosis, without being rejected, it will adhere to, and integrate with the local pubo-cervical fascia providing a fibrotic sheath, necessary for supporting and augmentation of the weak local fascia, and will be completely absorbed by the body

ELIGIBILITY:
Inclusion Criteria:

1 - Parity: from Para 1 to Para 5. 2-BMI: from 25 to 35 KG/M².

Exclusion Criteria:

1. Chronic debilitating diseases.
2. Conditions that lead to increase intra-abdominal pressure

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Awareness of prolapse and repair | From baseline to 3 months after the repair of vaginal prolapse operration
  Significant improvement of dyspareunia postoperative in patients with surgical repair of vaginal wall prolapse using Gamma Irradiated Amniotic Membrane

CONTACTS AND LOCATIONS:
Locations (1):
- SAYED GALAL HOSPITAL, AND AlGalaaTeaching HOSPITAL, Cairo, Egypt